CLINICAL TRIAL: NCT07367945
Title: Effect of Incentive Spirometry Versus Inspiratory Muscle Training on Arterial Blood Gases After Coronary Artery Bypass Grafting
Brief Title: Incentive Spirometry Versus Inspiratory Muscle Training After Coronary Artery Bypass Grafting
Acronym: IS/ IMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Abdelmohsen Ismail Hassan, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006065
Record Dates: First submitted 2026-01-06; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Bypass Graft (CABG)
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IS (Experimental): This group will include 15 patients, Incentive spirometry was utilized by the patient with ten breaths, six sets per day for a period of 10 min within patient tolerance in every session for five days with routinely physical therapy program (education and explanation) preoperatively, And postoperatively treatment (breathing treatment, deep-breathing applications, guided coughing, early mobilization).
  Interventions: Device: Incentive spirometry
- IMT (Experimental): This group will include 15 patients, each session consisted of 30 minutes of inspiratory muscle training. The patients were trained to use an inspiratory threshold-loading device (Threshold Inspiratory Muscle Training) for five days with routinely physical therapy program (education and explanation) preoperatively, And postoperatively treatment (breathing treatment, deep-breathing applications, guided coughing, early mobilization).
  Interventions: Device: Inspiratory muscle trainer
- Control group (Active Comparator): 15 patients will receive for 5 days routinely physical therapy program (education and explanation) preoperatively, And postoperatively treatment (breathing treatment, deep-breathing applications, guided coughing, early mobilization).
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Device: Incentive spirometry — This group will include 15 patients, Incentive spirometry was utilized by the patient with ten breaths, six sets per day for a period of 10 min within patient tolerance in every session for five days with routinely physical therapy program (education and explanation) preoperatively, And postoperatively treatment (breathing treatment, deep-breathing applications, guided coughing, early mobilization).
  Other Names: IS
  Arms: IS
Device: Inspiratory muscle trainer — This group will include 15 patients, each session consisted of 30 minutes of inspiratory muscle training. The patients were trained to use an inspiratory threshold-loading device (Threshold Inspiratory Muscle Training) for five days with routinely physical therapy program (education and explanation) preoperatively, And postoperatively treatment (breathing treatment, deep-breathing applications, guided coughing, early mobilization).
  Other Names: IMT
  Arms: IMT
Other: Routine physical therapy — 15 patients will receive for 5 days routinely physical therapy program (education and explanation) preoperatively, And postoperatively treatment (breathing treatment, deep-breathing applications, guided coughing, early mobilization).
  Other Names: Control group
  Arms: Control group

SUMMARY:
This study will be conducted to compare between incentive spirometry verses inspiratory muscle training preoperatively on (ABG) after coronary artery bypass graft surgery.

Is there any significant difference of preoperative incentive spirometry verses inspiratory muscle training on Arterial blood gases (ABG) after coronary artery bypass graft surgery?

Participants will:

Group A (incentive spirometry group ) Group B (Inspiratory muscle trainer group ) for 5 days before operative Group C (control group) and group a , b will have routinely postoperative

ELIGIBILITY:
Inclusion Criteria:

* 45 male patients will be included in this study.
* Patients with age from 50 to 60 years old (undergoing coronary artery bypass graft surgery) through median sternotomy.
* Their body mass index from 25 to 29.9 kg/m2
* Patients will be alert and able to follow instruction.

Exclusion Criteria:

* Who are expected not to be able to conduct or comply with IS and IMT.
* Patients with cognitive or neurological deficits.
* Patients with coexisting acute or chronic respiratory disorders.
* Patients unable to understand or show the proper use of the incentive spirometer and Inspiratory muscle training .
* Patients who cannot be instructed or supervised to assure appropriate use of the device patients in whom cooperation is absent or patients unable to understand or demonstrate proper use of the devices (inspiratory muscle training and incentive spirometry).
* Patients who are confused or delirious.
* Patients undergoing any other surgery along with CABG.
* Patients undergoing emergency CABG surgery.
* Chronic obstructive pulmonary disease (COPD), asthma, restrictive lung disease, preoperative major chest infection e.g. pulmonary tuberculosis, chest deformities such as pectus carinatum, pectus excavatum, thoracolumbar scoliosis, diaphragmatic hernias diagnosed on history.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Arterial Blood gas Parameters (PaO2 and SaO2) | Baseline 5 days pre-surgery , Immediately after the surgery within 48 hours , and through study completion an average of 8 days.
  Assessment of arterial oxygenation changes by measuring PaO2 and SaO2 . data will be collected at Baseline pre-surgery (5 days ) , Immediately after the surgery (within 48 hours) , and through study completion an average of 8 days.to evaluate the recovery trend and the effectiveness of respiratory interventions.

SECONDARY OUTCOMES:
Atelactasis | Baseline 5 days pre-surgery, Immediately after the surgery within 48 hours, and through study completion an average of 8 days.
  Assessment of lung collapse using chest X-ray and CT or clinical findings.
Functional capacity (2- minute walk test) | Baseline 5 days pre-surgery, and through study completion an average of 8 days.
  measuring the maximum distance a patient can walk on a flat surface in 2-minutes to evaluate functional exercise capacity.
Physical function ICU test - scored (PFIT-s) | Immediately after the surgery within 48 hours.
  Assessment of physical function in the ICU through four components ( sit -to- stand, marching, shoulder flexion, and knee extension ) Scored (0 - 10).
Mechanical Ventilation duration | from the end of surgery until successful extubation .
  the total number of hours the patient required mechanical ventilation support after CABG surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Alsharqia, Egypt

IPD SHARING:
Plan to Share IPD: No
data is available with a corresponding offer on reasonable request